CLINICAL TRIAL: NCT05505162
Title: An Open-Label, Single-Sequence Study to Assess the Effect of Multiple Doses of Zibotentan on the Pharmacokinetics of Single Doses of Combined Oral Ethinyl Estradiol and Levonorgestrel in Healthy Female Participants of Non-Child-Bearing Potential
Brief Title: Assessing the Effect of Multiple Doses of Zibotentan on the Pharmacokinetics of Single Doses of Combined Oral Contraceptives in Healthy Female Participants of Non-childbearing Potential.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4325C00006
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy Female Participants
Keywords: Ethinyl estradiol; Levonorgestrel; Zibotentan; Chronic Kidney Disease; Non-Child-Bearing Potential; Drug-drug interaction
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zibotentan and EE/LNG (Experimental): Participants will receive two tablets of combined oral EE/LNG on Day 1 with PK samples obtained from pre-dose on Day 1 until post-dose on Day 6.
  Participants will receive two capsules of zibotentan orally QD from Day 6 to Day 14. From Day 15 until Day 19 participants will continue to receive two capsules of zibotentan QD administered orally.
  On Day 15, participants will receive two tablets of combined oral EE and LNG with PK samples obtained pre-dose on Day 15 until post-dose (Day 20).
  Interventions: Drug: Zibotentan; Drug: EE/LNG

INTERVENTIONS:
Drug: Zibotentan — Participants will receive two capsules of Zibotentan orally QD from day 6-19.
Drug: EE/LNG — Participants will receive two tablets of EE and LNG once on Day 1 and Day 15 as a combined oral dose.

SUMMARY:
A study to assess the Pharmacokinetics (PK) of combined oral ethinyl estradiol (EE) and levonorgestrel (LNG) in healthy female participants of non-child-bearing potential, when administered alone and in combination with multiple oral doses of zibotentan.

DETAILED DESCRIPTION:
This is an open-label, single-sequence study conducted at a single study center.

The study will comprise of the following:

* A Screening Period (Visit 1) of maximum 28 days (Day -28 to Day -2).
* Treatment Period 1/Day 1 to Day 5 (in-house stay): Participants will check in at the clinical unit on Day -1 and will be resident at the clinical unit until Day 6.
* Treatment Period 2/Day 6 to Day 14 (home): Outpatient period.
* Treatment Period 3/Day 15 to Day 20 (in-house stay): On the evening of Day 14, the participants will check in at the clinical unit and will be resident at the clinical unit until Day 20.
* A follow-up visit (Day 27) will be conducted 7 days (±2 days) after the last PK sample collection (120 hours post-dose [Day 20]).

Participants will receive two tablets of EE/LNG on days 1 and 15 and 2 capsules of zibotentan on days 6-19.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the protocol.
* Healthy female participants aged 35 to 75 years (inclusive) at Day -1 with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and within 24 hours prior to dosing with EE/LNG on Day 1 and Day 15, must not be lactating and must be of non childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  (i) Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range [FSH > 40 mIU/mL].

(ii) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

* Have a body mass index (BMI) between 18.5 and 35 kg/m2 inclusive at Day -1.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study. Clinically significant diseases or disorders also include, but are not limited to:

  (i) Undiagnosed abnormal uterine bleeding, (ii) Current diagnosis of, or history of breast cancer, which may be hormone sensitive, (iii) Liver tumors, benign or malignant, or liver disease. Acute viral hepatitis, or severe (decompensated) cirrhosis or use of hepatitis C drug combinations containing ombitasvir/paritaprevir/ritonavir, with or without dasabuvir, due to the potential for alanine aminotransferase (ALT) elevations.
* Sex hormone therapy within 1 month before study.
* Current diagnosis or history of arterial or venous thrombosis (eg, deep vein thrombosis (DVT), pulmonary embolism (PE)), or known heredity risk factors (eg, activated protein C resistance), or coronary artery disease.
* Have inherited or acquired hypercoagulopathy.
* Participants treated with strong or moderate Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 3 months or longer (5 half-lives) prior to first administration of IMP in this study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any laboratory values with the following deviations:

  (i) Alanine aminotransferase > Upper limit of normal (ULN) (ii) Aspartate aminotransferase > ULN (iii) estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 (iv) Creatinine > 1.5 ULN (v) White blood cell count < 3.5 x 109/L (vi) Hemoglobin < lower limit of normal (LLN)
* Prolonged QT interval (QTcF > 470 ms) on ECG at check in into the clinical unit on Day 1 of Treatment Period 1, known congenital long QT syndrome or history of QT prolongation associated with other medications.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to zibotentan.
* Participants who have received zibotentan within 1 month prior to Day 1 dosing.
* Any of the following signs or confirmation of COVID-19 infection:

  (i) Positive COVID-19 test result on check in into the clinical unit on Day -1 and on Day 14.

(ii) Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnoea, sore throat, and fatigue) on check in into the clinical unit on Day 1.

(iii) Previously hospitalized with COVID-19 infection within the last 3 months prior to the screening visit.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are recruited
Enrollment: 24 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Terminal elimination half-life (t1/2λz) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Time to reach maximum observed concentration (tmax) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Apparent total body clearance of drug from plasma (CL/F) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.
Apparent volume of distribution based on terminal phase (Vz/F) | Day 1 and Day 15
  The effect of multiple doses of zibotentan on the PK of a single dose of combined oral EE and LNG in healthy female volunteers of non-child-bearing potential will be assessed.

SECONDARY OUTCOMES:
Area under plasma concentration-time curve in the dose interval (AUCtau) | Day 15
  The PK of zibotentan in healthy female volunteers of non-child-bearing potential will be assessed.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 15
  The PK of zibotentan in healthy female volunteers of non-child-bearing potential will be assessed.
Time to reach maximum observed concentration (tmax) | Day 15
  The PK of zibotentan in healthy female volunteers of non-child-bearing potential will be assessed.
Number of participants with adverse events | Until Follow up visit (7 days +/-2 days after last PK sample)
  The safety and tolerability of zibotentan alone and in combination with combined oral EE and LNG will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home